CLINICAL TRIAL: NCT01285804
Title: Impact of Using a Cuffed Endotracheal Tube on Limiting the Risk of Airway Fire
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chairman Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB10-00487
Record Dates: First submitted 2011-01-26; First posted 2011-01-28 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Adenoidectomy; Tonsillectomy; Adenotonsillectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cuffed ETT (Active Comparator)
  Interventions: Other: Cuffed ETT
- Uncuffed ETT (Active Comparator)
  Interventions: Other: Uncuffed ETT

INTERVENTIONS:
Other: Cuffed ETT — Kimberly Clark
  Arms: Cuffed ETT
Other: Uncuffed ETT — Kimberly Clark
  Arms: Uncuffed ETT

SUMMARY:
The purpose of this study is to evaluate the impact of using a cuffed endotracheal tube (ETT) on the oxygen concentration in the oropharynx during adenoidectomy, tonsillectomy, or adenotonsillectomy. The study hypothesis is that inflation of the cuff on the ETT will eliminate contamination of the oropharynx with the inspired anesthetic gases and decrease the oxygen concentration in the oropharynx.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing adenoidectomy, tonsillectomy, or adenotonsillectomy.

Exclusion Criteria:

* Airway anomalies or cardiac conditions that have the potential for a complicated anesthesia induction.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Difference in oxygen concentration in the oropharynx between cuffed and uncuffed ETT. | 4-5 minutes after induction
  The oxygen and sevoflurane (anesthetic agent) concentration of the oropharynx would be measured during positive pressure ventilation immediately after intubation and then 4-5 mins. after anesthetic induction when the patient resumes spontaneous ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States